CLINICAL TRIAL: NCT03295877
Title: A Phase I, Multicenter, Open-Label, Single-Dose, Dose-Escalation, and Multiple-Dose Study of the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of Intravitreal Injections of RO7171009 in Patients With Geographic Atrophy Secondary to Age-Related Macular Degeneration
Brief Title: Safety and Tolerability Study of RO7171009 in Participants With Geographic Atrophy (GA) Secondary to Age-Related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GR39821
Record Dates: First submitted 2017-09-19; First posted 2017-09-28 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RO7171009: SAD (Experimental): Patients will receive a single dose of RO7171009, in multiple escalating cohorts.
  Interventions: Drug: RO7171009
- RO7171009: MD (Experimental): Patients will receive RO7171009 at maximum tolerated dose (MTD), identified during the SAD stage for three doses.
  Interventions: Drug: RO7171009

INTERVENTIONS:
Drug: RO7171009 — Patients will receive RO7171009 via ITV injection.

SUMMARY:
This Phase 1, open-label, multicenter study will investigate the safety and tolerability of RO7171009 following single and multiple intravitreal (ITV) administrations in patients with GA secondary to AMD. The study consists of two stages: Single Dose-Escalation (SAD) and Multiple-Dose (MD) stages.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged greater than or equal to (>/=) 50 years
* Well demarcated area(s) of GA secondary to AMD with no evidence of prior or active choroidal neovascularization (CNV) in study eye

Exclusion Criteria:

Ocular Exclusion Criteria, Study Eye:

* History of vitrectomy surgery, submacular surgery, or other surgical intervention for AMD
* Previous laser photocoagulation for CNV, diabetic macular edema, retinal vein occlusion, or proliferative diabetic retinopathy
* Prior treatment with Visudyne®, external beam radiation therapy (for intraocular conditions), or transpupillary thermotherapy

Ocular Exclusion Criteria (Both Eyes):

* GA in either eye due to causes other than AMD
* Evidence of prior or active CNV
* Previous participation in interventional clinical trials for GA or dry AMD, except for vitamins and minerals, irrespective of the route of administration (i.e., ocular or systemic) within the last 6 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of the Study Drug: Rate of Adverse Events | Through study completion or early study discontinuation (overall 12-20 weeks)

SECONDARY OUTCOMES:
Serum Concentration of RO7171009 | Through study completion or early study discontinuation (overall 12-20 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- United States (13):
  - California Retina Consultants, Bakersfield, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Retinal Consultants Med Group, Sacramento, California
  - California Retina Consultants, Santa Barbara, California
  - California Retina Consultants - Santa Maria, Santa Maria, California
  - Retina Consultants of Southern Colorado PC; Clinical Research Department, Colorado Springs, Colorado
  - Florida Eye Associates, Melbourne, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Georgia Retina PC, Marietta, Georgia
  - The Retina Institute, St Louis, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - Western Carolina Retinal Associate PA, Asheville, North Carolina
  - Tennessee Retina PC., Nashville, Tennessee